CLINICAL TRIAL: NCT00790114
Title: A Phase I Open-Labeled, Fixed Sequence Study to Determine the Effect of Multiple Doses of AZD7325 on the Pharmacokinetics of Midazolam (CYP3A4) and Caffeine (CYP1A2)
Brief Title: Determine the Effect of Multiple Doses of AZD7325, CYP Study
Acronym: CYP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark A. Smith, MD, PhDMedical Science Sr.Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: D1140C00005
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Healthy Volunteer
Keywords: Phase I
MeSH Terms: interventions — 4-amino-8-(2-fluoro-6-methoxy-phenyl)-N-propylcinnoline-3-carboxamide; Midazolam; Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD7325; Drug: Midazolam; Drug: Caffeine

INTERVENTIONS:
Drug: AZD7325 — Oral, day 1-12
Drug: Midazolam — single dose, twice during treatment
Drug: Caffeine — single dose, twice during treatment

SUMMARY:
To determine the effects of repeated doses of AZD7325 on the pharmacokinetic profile of a CYP3A4 substrate (midazolam and its 1' hydroxy metabolite) and a CYP1A2 substrate (caffeine and its paraxanthine [3-desmethyl] metabolite).

ELIGIBILITY:
Exclusion Criteria:

* Clinically relevant abnormalities in physical examinations, vital signs, clinical chemistry, hematology or urinalysis as judged by the investigator and/or sponsor.
* Enrollment in another concurrent investigational study or intake of an investigational drug within 3 months or intake of an investigational drug within a period of 5 half lives of that drug prior to the screening visit

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To determine the effects of repeated doses of AZD7325 on the pharmacokinetic profile of a CYP3A4 substrate (midazolam and its 1' hydroxy metabolite) and a CYP1A2 substrate (caffeine and its paraxanthine [3-desmethyl] metabolite). | Blood samples will be taken during the study.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of repeated doses of AZD7325 in combination with midazolam and caffeine. | Blood samples will be taken during the study.
Evaluation of the pharmacodynamic effects of AZD7325 | Test batteries will be performed at specified times both before and following study drug administration.
To evaluate the pharmacokinetics of AZD7325 | Blood samples will be taken on Days 1, 11 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MBBS, DCPSA, Principal Investigator — Guy's Drug Research Unit Quintiles